CLINICAL TRIAL: NCT03725631
Title: Non-invasive Evaluation of Liver Fibrosis, Steatosis, and Nonalcoholic Steatohepatitis in Biopsy-Proven NAFLD Patients
Brief Title: Non-invasive Evaluation of Liver Fibrosis, Steatosis, and NASH in NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Jong Eun Yeon, Professor, Korea University Guro Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016GR0302
Record Dates: First submitted 2018-08-20; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis
Keywords: Magnetic resonance imager(MRI); Nonalcoholic fatty liver disease(NAFLD); Biomarker
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy proven NAFLD patients (Experimental): 150 subjects who are diagnosed with NAFLD with biopsy from September 2016 to October 2018.
  Interventions: Diagnostic Test: Imaging and serologic evaluation of fibrosis and steatosis

INTERVENTIONS:
Diagnostic Test: Imaging and serologic evaluation of fibrosis and steatosis — Imaging evaluation: Fibroscan, MRI scan for evaluation of fibrosis and steatosis in biopsy proven NAFLD patients Serologic evaluation: serologic test for evaluation of fibrosis and steatosis in biopsy proven NAFLD patients

SUMMARY:
1. To evaluate hepatic fibrosis and steatosis using MR imaging, transient elastography (TE), and serum biomarker
2. To develop non-invasive diagnosis marker for NASH and advanced fibrosis

DETAILED DESCRIPTION:
As nonalcoholic fatty liver disease (NAFLD) is becoming a leading cause of chronic liver disease, non-invasive diagnosis of disease severity in NAFLD is urgently needed. In this study, the investigators compared hepatic fibrosis and steatosis using MR imaging and transient elastography (TE) and tried to find non-invasive diagnostic marker for NASH and advanced fibrosis.

This is a multicenter prospective study of patients with biopsy-proven NAFLD. The patients were underwent laboratory test, liver biopsy, MRI and TE within 6 months of enrollment. MRI examination included MR spectroscopy (MRS), and MR elastography (MRE). TE measured liver stiffness and controlled attenuation parameter (CAP).

ELIGIBILITY:
Inclusion Criteria:

* Patients >19 years age
* Patients who had elevated aspartate transaminase(AST)/alanine transaminase(ALT) or fatty liver on abdominal ultrasonography
* Patients who are clinically suspected to have nonalcoholic steatohepatitis(NASH): >40 years age, BMI >25, multiple features of the metabolic syndrome, presence of diabetes mellitus (DM) , fibroscan > 6 kilopascal (kPa), platelet count < 150,000 /ml, and other patients suspected to progress clinically or requiring diagnosis
* Patients who underwent (<6 months) or will undergo US-guided liver biopsy

Exclusion Criteria:

* Chronic liver disease other than nonalcoholic fatty liver disease(NAFLD) (chronic hepatitis B or C, autoimmune hepatitis, primary biliary cholangitis)
* Excessive alcohol consumption (weekly men >140g and women >70g)
* Fatty liver due to medication
* Decompensated liver cirrhosis
* Contraindication to magnetic resonance imager(MRI)
* Malignancy or other systemic disease
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Development of scoring system for diagnosis of NASH | up to 24 months
  Development of scoring system for diagnosis of NASH using cox regression analysis

SECONDARY OUTCOMES:
Evaluation of hepatic fibrosis using fibroscan | up to 24 months
  Assessment of hepatic fibrosis using fibroscan with transient elastography (kilopascals) (kPa)
Evaluation of hepatic steatosis using fibroscan | up to 24 months
  Assessment of hepatic steatosis using fibroscan with CAP (Controlled Attenuation Parameter) (dB/m)
Evaluation of hepatic fibrosis using MRI | up to 24 months
  Assessment of hepatic fibrosis using MRI with MR elastography (MRE) (kPa)
Evaluation of hepatic steatosis using MRS | up to 24 months
  Assessment of hepatic steatosis using fibroscan with MR spectrography (MRS) (%)
Evaluation of hepatic fibrosis using serologic marker | up to 24 months
  Assessment of hepatic fibrosis using AST to Platelet Ratio Index (APRI)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Eun Yeon, MD, Ph.D., Principal Investigator — Prefessor
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-23. doi: 10.1002/hep.25762. No abstract available. PMID 22488764
- [Background] Poynard T, Lenaour G, Vaillant JC, Capron F, Munteanu M, Eyraud D, Ngo Y, M'Kada H, Ratziu V, Hannoun L, Charlotte F. Liver biopsy analysis has a low level of performance for diagnosis of intermediate stages of fibrosis. Clin Gastroenterol Hepatol. 2012 Jun;10(6):657-63.e7. doi: 10.1016/j.cgh.2012.01.023. Epub 2012 Feb 14. PMID 22343514
- [Background] Banerjee R, Pavlides M, Tunnicliffe EM, Piechnik SK, Sarania N, Philips R, Collier JD, Booth JC, Schneider JE, Wang LM, Delaney DW, Fleming KA, Robson MD, Barnes E, Neubauer S. Multiparametric magnetic resonance for the non-invasive diagnosis of liver disease. J Hepatol. 2014 Jan;60(1):69-77. doi: 10.1016/j.jhep.2013.09.002. Epub 2013 Sep 12. PMID 24036007
- [Background] Park YS, Lee CH, Kim JH, Kim BH, Kim JH, Kim KA, Park CM. Effect of Gd-EOB-DTPA on hepatic fat quantification using high-speed T2-corrected multi-echo acquisition in (1)H MR spectroscopy. Magn Reson Imaging. 2014 Sep;32(7):886-90. doi: 10.1016/j.mri.2014.04.010. Epub 2014 Apr 24. PMID 24853467
- [Background] Ishak K, Baptista A, Bianchi L, Callea F, De Groote J, Gudat F, Denk H, Desmet V, Korb G, MacSween RN, et al. Histological grading and staging of chronic hepatitis. J Hepatol. 1995 Jun;22(6):696-9. doi: 10.1016/0168-8278(95)80226-6. No abstract available. PMID 7560864
- [Background] Brunt EM, Janney CG, Di Bisceglie AM, Neuschwander-Tetri BA, Bacon BR. Nonalcoholic steatohepatitis: a proposal for grading and staging the histological lesions. Am J Gastroenterol. 1999 Sep;94(9):2467-74. doi: 10.1111/j.1572-0241.1999.01377.x. PMID 10484010
- [Background] SCHEUER PJ, WILLIAMS R, MUIR AR. Hepatic pathology in relatives of patients with haemochromatosis. J Pathol Bacteriol. 1962 Jul;84:53-64. No abstract available. PMID 14498313
- [Background] Kleiner DE, Brunt EM, Van Natta M, Behling C, Contos MJ, Cummings OW, Ferrell LD, Liu YC, Torbenson MS, Unalp-Arida A, Yeh M, McCullough AJ, Sanyal AJ; Nonalcoholic Steatohepatitis Clinical Research Network. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology. 2005 Jun;41(6):1313-21. doi: 10.1002/hep.20701. PMID 15915461
- [Background] Piechnik SK, Ferreira VM, Dall'Armellina E, Cochlin LE, Greiser A, Neubauer S, Robson MD. Shortened Modified Look-Locker Inversion recovery (ShMOLLI) for clinical myocardial T1-mapping at 1.5 and 3 T within a 9 heartbeat breathhold. J Cardiovasc Magn Reson. 2010 Nov 19;12(1):69. doi: 10.1186/1532-429X-12-69. PMID 21092095